CLINICAL TRIAL: NCT05985226
Title: Clinical Evaluation of the Effect of the Scanning Pattern on Complete-arch Implant Scans
Acronym: strategiesIOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C.I. 22/645-E
Record Dates: First submitted 2023-07-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-11

CONDITIONS: Dental Prosthesis, Implant-Supported
Keywords: Accuracy; intraoral scanners; digital impressions; complete arch; implant-supported dental prostheses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- scanning strategies (Experimental): 6 experimental groups will be created based on the strategy-scan body used (1.- zigzag with conventional scan body (ZZ-SBL), 2.- circumferential with conventional scan body (C-SBL), 3.- surface blocking with scan conventional body (B-SBL), 4.- zigzag with low profile scan body (ZZ-SBL), 5.- a standard strategy with low profile scan body (STD-SBL), 6.- single pass with low profile scan body ( OP-SBL) These experimental groups will be scanned directly in the patient's mouth, to later be compared with the reference model, called the "master model".
  Interventions: Device: intraoral scan

INTERVENTIONS:
Device: intraoral scan — All the experimental groups will be developed with an intraoral scanner, a device that emits light and collects the image projected by that light, to build a 3-dimensional digital model. It is more comfortable than conventional impressions and it is a harmless, non-intrusive, and painless procedure.

SUMMARY:
This clinical trial aims to analyze and compare the influence of different scanning strategies (zigzag with conventional scan body, circumferential with conventional scan body, surface blocking with conventional scan body, zigzag with low profile scan body, standard strategy with low profile scan body) on the accuracy of the records obtained for a case of fixed rehabilitation on full-arch dental implants in patients of both sexes, over 18 years of age who will be rehabilitated with fixed prostheses on full-arch implants.

The main question it aims to answer is if there will be significant differences in scanning accuracy (trueness and precision) between the different groups of digital impressions compared to the reference model (conventional impression with rigid splinting) and types of scan bodies.

The patient will undergo conventional impression-taking (with pastes) to obtain the reference model. Subsequently, digital records will be taken with the intra-oral scanner until completing 15 records per group, out of a total of 6 experimental groups (1.- zigzag with conventional scan body (ZZ-SBL), 2.- circumferential with conventional scan body (C-SBL), 3.- surface blocking with scan conventional body (B-SBL), 4.- zigzag with low profile scan body (ZZ-SBL), 5.- a standard strategy with low profile scan body (STD-SBL), 6.- single pass with low profile scan body ( OP-SBL) These experimental groups will be scanned directly in the patient's mouth, to later be compared with the reference model, called the "master model".

Researchers will compare the six different methodologies for taking digital impressions to demonstrate which strategies are more accurate, faster, and require fewer frames.

DETAILED DESCRIPTION:
INTRODUCTION AND BACKGROUND Record-taking is a fundamental process and the starting point for manufacturing a dental prosthesis. The appearance of intraoral scanners (IntraOral Scanners (IOS)) has meant a revolution in this regard due to the advantages they provide, including better communication with both the patient and the dental laboratory, better comfort and acceptance by the patient, the immediacy in sending the file and saving space in the storage of digital models versus conventional ones. However, they are not exempt from problems, including their high cost, the learning curve, and difficulty achieving a reliable record in certain circumstances, including edentulous full-arch records.

Recordings of the edentulous full arch with IOSs pose a challenge due to the type of operation of these devices, which gradually collect and overlap information from small areas until completing a full arch. For this reason, different techniques have been proposed to improve the accuracy of this type of recording. In addition, if there is a case in which accuracy is crucial, it is complete edentulous arches with implants since, if the registration is not exact, the prosthesis manufactured on it will not have a passive fit in the mouth, which would lead to the appearance of both biological and mechanical complications.

Different studies have tried to analyze how various factors influence this accuracy, and these factors can be divided into factors related to the operator, the scanner, environmental conditions, or intraoral conditions-also different scanning strategies or heights and positions of the scan bodies. However, most of these works have been developed in an in vitro environment. This fact is motivated by the greater ease of making the records and, as a more relevant fact, the possibility of obtaining a reliable reference model, employing a coordinate machine (Coordinate Measurement Machine (CMM)) or a desktop scanner, something that in an in vivo study it is not possible.

The present study aims to clinically analyze the accuracy of different intraoral scanning strategies and types of scan bodies in edentulous full arch registrations on implants.

JUSTIFICATION Due to the importance of the accuracy in taking digital impressions in full-arch patients for the fabrication of restorations on implants, it is considered justified to study the influence of different scanning strategies and scan bodies on the accuracy of full-arch recording.

VIABILITY The project could be considered viable by having all the instruments and apparatus necessary to develop the material and methods. It is estimated that the proposed methodology could be developed within the period described.

AIM The purpose of this in vivo study will be to measure the influence of different scanning strategies (zigzag with conventional scan body, circumferential with conventional scan body, surface blocking with conventional scan body, zigzag with low profile scan body, standard strategy with low profile scan body) on the accuracy of the records obtained for a case of fixed rehabilitation on full-arch dental implants.

HYPOTHESIS The null hypothesis will be that there are no significant differences in scanning accuracy (trueness and precision) between the different groups of digital impressions compared to the reference model (conventional impression with rigid splinting).

The alternative hypothesis will be that there are significant differences in scanning accuracy (trueness and precision) between the different groups of digital impressions compared to the reference model (conventional impression with rigid splinting).

MATERIAL AND METHOD A patient will be selected who is susceptible to rehabilitation with a fixed prosthesis on implants, in good general health (ASA I and ASA II), without joint problems or limitation of opening, and who, after reading the information sheet, the patient and informed consent, and clarified any doubts, voluntarily agree to participate in the study.

A reference model will be taken with a high-precision conventional methodology such as Rigid Impression Splinting. A first impression will be taken with double-mix addition silicone (putty and fluid) with an open tray. From this record, a first model will be generated that will be used to splint the impression transfers with a rigid, low-shrinkage light-curing material, which will later be sectioned with discs. Subsequently, the transfers will be screwed with the splint in the mouth and rejoined using a low-shrinkage light-curing material, thus minimizing the possibility of accumulation of errors. A second impression will be taken dragging the entire set, and it will be cast in improved type IV plaster (GC Fujirock; GC), thus obtaining the master model. This model will be digitized using a laboratory scanner to get the reference digital model, against which the specimens resulting from the experimental groups will be compared.

Six experimental groups will be created based on the strategy-scan body used (1.- zigzag with conventional scan body (ZZ-SBL), 2.- circumferential with conventional scan body (C-SBL), 3.- surface blocking with scan conventional body (B-SBL), 4.- zigzag with low profile scan body (ZZ-SBL), 5.- a standard strategy with low profile scan body (STD-SBL), 6.- single pass with low profile scan body ( OP-SBL) These experimental groups will be scanned directly in the patient's mouth, to be compared with the reference model, called the "master model".

Based on previous studies, a sample size of n=15 is estimated for each group. A pilot study will be carried out with n=5, from which a statistical test (G* Power; University of Düsseldorf) will be carried out to calculate the sample size. All digitization procedures will be performed under lighting conditions of 1000 lux measured with a lux meter (LX1330B Light Meter; Dr. Meter Digital Illuminance) and at a constant temperature of 24 +/-2 ºC. Once the files are obtained, they will be exported with the reference format for a 3-dimensional.STL (standard tessellation language) file to a metrology program (Geomagic Control X). The results will be compared with a reference file, and the deviations of the implant positions will be obtained using the best-fit algorithm. The mean square error (Root Mean Square) will be calculated.

statistical plan Statistical tests will be developed to check the normal distribution of the samples, Shapiro-Wilk or Kolmogorov-Smirnov type. A priori tests will be carried out to verify the existence of statistically significant differences, and a posteriori for analyzing which groups such differences appear and their magnitude. Statistical power will be 95%, so those with p<.05 will be considered statistically significant differences. All statistical analysis will be performed using a statistical software program (IBM SPSS Statistics for Windows, v26; IBM Corp).

VARIABLES COLLECTED AND DESCRIPTION OF THE ACTIONS TO BE CARRIED OUT AND FINAL DESTINATION OF THE SAMPLES The collected variable is the discrepancy in the position of the implants between the control model, reference, and the experimental groups, quantified as a Root Mean Square. The samples, in this case, files, will be saved anonymously on a hard drive, named so that the group to which they belong and the number of samples can be interpreted (Example: ZZ-SBL1). The scanning time and the number of frames will also be collected.

SCHEDULE December 2022-March 2023: collection, sample preparation, development of experimental methodology, and data collection.

April 2023-July 2023: Statistical analysis and writing of the manuscript.

ETHICAL IMPLICATIONS To the best of the research team's knowledge, the most significant ethical implication lies in carrying out several recordings of the same patient. In this regard, it should be noted that, in addition to meeting the inclusion requirements, the participant wishes to participate completely voluntarily and know that the participant will not obtain any compensation, financial or in any other way. On the other hand, we must bear in mind that intraoral record-taking procedures with intraoral scanners can be considered harmless and painless, which simply means that the patient must keep his mouth open during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient susceptible to rehabilitation with a fixed prosthesis on implants.
* Good general health (ASA I and ASA II),

Exclusion Criteria:

* Joint problems or limitation of opening.
* Patients who, after reading the information sheet the patient and informed consent, and clarified any doubts, do not agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy | Up to 1 year
  Micrometers (root mean square deviations)

SECONDARY OUTCOMES:
Number of photograms | Up to 1 year
  Number of images
clinical scan time | Up to 1 year
  Seconds (s)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Gómez-Polo, PhD, DDS, Study Director — Universidad Complutense de Madrid
Locations (1):
- School of Dentistry, Complutense University. Pza Ramón y Cajal s/n., Madrid, Spain

REFERENCES:
- [Background] Gomez-Polo M, Cascos R, Ortega R, Barmak AB, Kois JC, Revilla-Leon M. Influence of arch location and scanning pattern on the scanning accuracy, scanning time, and number of photograms of complete-arch intraoral digital implant scans. Clin Oral Implants Res. 2023 Jun;34(6):591-601. doi: 10.1111/clr.14069. Epub 2023 Apr 13. PMID 37052054
- [Background] Zhang YJ, Shi JY, Qian SJ, Qiao SC, Lai HC. Accuracy of full-arch digital implant impressions taken using intraoral scanners and related variables: A systematic review. Int J Oral Implantol (Berl). 2021 May 12;14(2):157-179. PMID 34006079
- [Background] Rignon-Bret C, Wulfman C, Hadida A, Renouard F, Gourraud PA, Naveau A. Immediate Loading of Two Unsplinted Implants in Edentulous Patients with Mandibular Overdentures: A 10-year Retrospective Review of Patients from a Previously Conducted 1-year Cohort Study. Int J Oral Maxillofac Implants. 2019 Jan/Feb;34(1):169-178. doi: 10.11607/jomi.6931. PMID 30695092
- [Background] Tabesh M, Nejatidanesh F, Savabi G, Davoudi A, Savabi O. Marginal Accuracy of Lithium Disilicate Full-Coverage Single Crowns Made by Direct and Indirect Digital or Conventional Workflows: A Systematic Review and Meta-Analysis. J Prosthodont. 2022 Dec;31(9):744-753. doi: 10.1111/jopr.13515. Epub 2022 May 10. PMID 35344238
- [Background] Schimmel M, Akino N, Srinivasan M, Wittneben JG, Yilmaz B, Abou-Ayash S. Accuracy of intraoral scanning in completely and partially edentulous maxillary and mandibular jaws: an in vitro analysis. Clin Oral Investig. 2021 Apr;25(4):1839-1847. doi: 10.1007/s00784-020-03486-z. Epub 2020 Aug 19. PMID 32812098
- [Background] Sallorenzo A, Gomez-Polo M. Comparative study of the accuracy of an implant intraoral scanner and that of a conventional intraoral scanner for complete-arch fixed dental prostheses. J Prosthet Dent. 2022 Nov;128(5):1009-1016. doi: 10.1016/j.prosdent.2021.01.032. Epub 2021 Apr 7. PMID 33836855
- [Background] Papaspyridakos P, Vazouras K, Chen YW, Kotina E, Natto Z, Kang K, Chochlidakis K. Digital vs Conventional Implant Impressions: A Systematic Review and Meta-Analysis. J Prosthodont. 2020 Oct;29(8):660-678. doi: 10.1111/jopr.13211. Epub 2020 Jul 16. PMID 32613641
- [Background] Revilla-Leon M, Gohil A, Barmak AB, Zandinejad A, Raigrodski AJ, Alonso Perez-Barquero J. Best-Fit Algorithm Influences on Virtual Casts' Alignment Discrepancies. J Prosthodont. 2023 Apr;32(4):331-339. doi: 10.1111/jopr.13537. Epub 2022 Jun 6. PMID 35524587
- [Background] Revilla-Leon M, Young K, Sicilia E, Cho SH, Kois JC. Influence of definitive and interim restorative materials and surface finishing on the scanning accuracy of an intraoral scanner. J Dent. 2022 May;120:104114. doi: 10.1016/j.jdent.2022.104114. Epub 2022 Mar 28. PMID 35358659
- [Background] Revilla-Leon M, Sicilia E, Agustin-Panadero R, Gomez-Polo M, Kois JC. Clinical evaluation of the effects of cutting off, overlapping, and rescanning procedures on intraoral scanning accuracy. J Prosthet Dent. 2023 Nov;130(5):746-754. doi: 10.1016/j.prosdent.2021.10.017. Epub 2022 Jan 6. PMID 34998582
- [Background] Revilla-Leon M, Gohil A, Barmak AB, Gomez-Polo M, Perez-Barquero JA, Att W, Kois JC. Influence of ambient temperature changes on intraoral scanning accuracy. J Prosthet Dent. 2023 Nov;130(5):755-760. doi: 10.1016/j.prosdent.2022.01.012. Epub 2022 Feb 21. PMID 35210107
- [Background] Revilla-Leon M, Quesada-Olmo N, Gomez-Polo M, Sicilia E, Farjas-Abadia M, Kois JC. Influence of rescanning mesh holes on the accuracy of an intraoral scanner: An in vivo study. J Dent. 2021 Dec;115:103851. doi: 10.1016/j.jdent.2021.103851. Epub 2021 Oct 15. PMID 34656658
- [Background] Revilla-Leon M, Subramanian SG, Att W, Krishnamurthy VR. Analysis of Different Illuminance of the Room Lighting Condition on the Accuracy (Trueness and Precision) of An Intraoral Scanner. J Prosthodont. 2021 Feb;30(2):157-162. doi: 10.1111/jopr.13276. Epub 2020 Nov 7. PMID 33094878
- [Background] Revilla-Leon M, Frazier K, da Costa JB, Kumar P, Duong ML, Khajotia S, Urquhart O; Council on Scientific Affairs. Intraoral scanners: An American Dental Association Clinical Evaluators Panel survey. J Am Dent Assoc. 2021 Aug;152(8):669-670.e2. doi: 10.1016/j.adaj.2021.05.018. PMID 34325781
- [Background] Revilla-Leon M, Subramanian SG, Ozcan M, Krishnamurthy VR. Clinical Study of the Influence of Ambient Lighting Conditions on the Mesh Quality of an Intraoral Scanner. J Prosthodont. 2020 Oct;29(8):651-655. doi: 10.1111/jopr.13205. Epub 2020 Jun 20. PMID 32463965
- [Background] Revilla-Leon M, Jiang P, Sadeghpour M, Piedra-Cascon W, Zandinejad A, Ozcan M, Krishnamurthy VR. Intraoral digital scans: Part 2-influence of ambient scanning light conditions on the mesh quality of different intraoral scanners. J Prosthet Dent. 2020 Nov;124(5):575-580. doi: 10.1016/j.prosdent.2019.06.004. Epub 2019 Dec 20. PMID 31870612
- [Background] Resende CCD, Barbosa TAQ, Moura GF, Tavares LDN, Rizzante FAP, George FM, Neves FDD, Mendonca G. Influence of operator experience, scanner type, and scan size on 3D scans. J Prosthet Dent. 2021 Feb;125(2):294-299. doi: 10.1016/j.prosdent.2019.12.011. Epub 2020 Feb 27. PMID 32115221
- [Background] Ren S, Jiang X, Lin Y, Di P. Crown Accuracy and Time Efficiency of Cement-Retained Implant-Supported Restorations in a Complete Digital Workflow: A Randomized Control Trial. J Prosthodont. 2022 Jun;31(5):405-411. doi: 10.1111/jopr.13447. Epub 2021 Dec 8. PMID 34748653
- [Background] Rasaie V, Abduo J, Falahchai M. Clinical and Laboratory Outcomes of Angled Screw Channel Implant Prostheses: A Systematic Review. Eur J Dent. 2022 Jul;16(3):488-499. doi: 10.1055/s-0041-1740298. Epub 2022 Feb 21. PMID 35189643
- [Background] Ochoa-Lopez G, Cascos R, Antonaya-Martin JL, Revilla-Leon M, Gomez-Polo M. Influence of ambient light conditions on the accuracy and scanning time of seven intraoral scanners in complete-arch implant scans. J Dent. 2022 Jun;121:104138. doi: 10.1016/j.jdent.2022.104138. Epub 2022 Apr 22. PMID 35461973
- [Background] Muller P, Ender A, Joda T, Katsoulis J. Impact of digital intraoral scan strategies on the impression accuracy using the TRIOS Pod scanner. Quintessence Int. 2016 Apr;47(4):343-9. doi: 10.3290/j.qi.a35524. PMID 26824085
- [Background] Morsy N, El Kateb M, Azer A, Fathalla S. Fit of zirconia fixed partial dentures fabricated from conventional impressions and digital scans: A systematic review and meta-analysis. J Prosthet Dent. 2023 Jul;130(1):28-34. doi: 10.1016/j.prosdent.2021.08.025. Epub 2021 Oct 23. PMID 34696907
- [Background] Moslemion M, Payaminia L, Jalali H, Alikhasi M. Do Type and Shape of Scan Bodies Affect Accuracy and Time of Digital Implant Impressions? Eur J Prosthodont Restor Dent. 2020 Feb 27;28(1):18-27. doi: 10.1922/EJPRD_1962Moslemion10. PMID 32036633
- [Background] Mizumoto RM, Jamjoom FZ, Yilmaz B. A risk-based decision making tree for managing fractured abutment and prosthetic screws: A systematic review. J Prosthet Dent. 2018 Apr;119(4):552-559. doi: 10.1016/j.prosdent.2017.05.016. Epub 2017 Sep 6. PMID 28888412
- [Background] Medina-Sotomayor P, Pascual-Moscardo A, Camps A I. Accuracy of 4 digital scanning systems on prepared teeth digitally isolated from a complete dental arch. J Prosthet Dent. 2019 May;121(5):811-820. doi: 10.1016/j.prosdent.2018.08.020. Epub 2018 Dec 28. PMID 30598308
- [Background] Imburgia M, Logozzo S, Hauschild U, Veronesi G, Mangano C, Mangano FG. Accuracy of four intraoral scanners in oral implantology: a comparative in vitro study. BMC Oral Health. 2017 Jun 2;17(1):92. doi: 10.1186/s12903-017-0383-4. PMID 28577366
- [Background] Lim JH, Mangal U, Nam NE, Choi SH, Shim JS, Kim JE. A Comparison of Accuracy of Different Dental Restorative Materials between Intraoral Scanning and Conventional Impression-Taking: An In Vitro Study. Materials (Basel). 2021 Apr 19;14(8):2060. doi: 10.3390/ma14082060. PMID 33921830
- [Background] Lim JH, Park JM, Kim M, Heo SJ, Myung JY. Comparison of digital intraoral scanner reproducibility and image trueness considering repetitive experience. J Prosthet Dent. 2018 Feb;119(2):225-232. doi: 10.1016/j.prosdent.2017.05.002. Epub 2017 Jul 8. PMID 28689906
- [Background] Lawand G, Ismail Y, Revilla-Leon M, Tohme H. Effect of implant scan body geometric modifications on the trueness and scanning time of complete arch intraoral implant digital scans: An in vitro study. J Prosthet Dent. 2024 Jun;131(6):1189-1197. doi: 10.1016/j.prosdent.2022.06.004. Epub 2022 Jul 19. PMID 35864021
- [Background] Kim MK, Son K, Yu BY, Lee KB. Effect of the volumetric dimensions of a complete arch on the accuracy of scanners. J Adv Prosthodont. 2020 Dec;12(6):361-368. doi: 10.4047/jap.2020.12.6.361. Epub 2020 Dec 28. PMID 33489020
- [Background] Park JM, Kim RJ, Lee KW. Comparative reproducibility analysis of 6 intraoral scanners used on complex intracoronal preparations. J Prosthet Dent. 2020 Jan;123(1):113-120. doi: 10.1016/j.prosdent.2018.10.025. Epub 2019 Apr 23. PMID 31027953
- [Background] Kaewbuasa N, Ongthiemsak C. Effect of different arch widths on the accuracy of three intraoral scanners. J Adv Prosthodont. 2021 Aug;13(4):205-215. doi: 10.4047/jap.2021.13.4.205. Epub 2021 Aug 26. PMID 34504672
- [Background] Jin-Young Kim R, Benic GI, Park JM. Trueness of intraoral scanners in digitizing specific locations at the margin and intaglio surfaces of intracoronal preparations. J Prosthet Dent. 2021 Dec;126(6):779-786. doi: 10.1016/j.prosdent.2020.09.019. Epub 2020 Nov 8. PMID 33176925
- [Background] Hasanzade M, Aminikhah M, Afrashtehfar KI, Alikhasi M. Marginal and internal adaptation of single crowns and fixed dental prostheses by using digital and conventional workflows: A systematic review and meta-analysis. J Prosthet Dent. 2021 Sep;126(3):360-368. doi: 10.1016/j.prosdent.2020.07.007. Epub 2020 Sep 12. PMID 32928518
- [Background] Gomez-Polo M, Sallorenzo A, Ortega R, Gomez-Polo C, Barmak AB, Att W, Revilla-Leon M. Influence of implant angulation and clinical implant scan body height on the accuracy of complete arch intraoral digital scans. J Prosthet Dent. 2024 Jan;131(1):119-127. doi: 10.1016/j.prosdent.2021.11.018. Epub 2022 Mar 23. PMID 35337658
- [Background] Gomez-Polo M, Alvarez F, Ortega R, Gomez-Polo C, Barmak AB, Kois JC, Revilla-Leon M. Influence of the implant scan body bevel location, implant angulation and position on intraoral scanning accuracy: An in vitro study. J Dent. 2022 Jun;121:104122. doi: 10.1016/j.jdent.2022.104122. Epub 2022 Apr 6. PMID 35395345
- [Background] Gomez-Polo M, Cimolai A, Ortega R, Barmak AB, Kois JC, Revilla-Leon M. Accuracy, scanning time, and number of photograms of various scanning patterns for the extraoral digitalization of complete dentures by using an intraoral scanner. J Prosthet Dent. 2024 Mar;131(3):521-528. doi: 10.1016/j.prosdent.2022.03.017. Epub 2022 May 5. PMID 35527066
- [Background] Gomez-Polo M, Piedra-Cascon W, Methani MM, Quesada-Olmo N, Farjas-Abadia M, Revilla-Leon M. Influence of rescanning mesh holes and stitching procedures on the complete-arch scanning accuracy of an intraoral scanner: An in vitro study. J Dent. 2021 Jul;110:103690. doi: 10.1016/j.jdent.2021.103690. Epub 2021 May 12. PMID 33991598
- [Background] Zimmermann M, Ender A, Attin T, Mehl A. Fracture load of three-unit full-contour fixed dental prostheses fabricated with subtractive and additive CAD/CAM technology. Clin Oral Investig. 2020 Feb;24(2):1035-1042. doi: 10.1007/s00784-019-03000-0. Epub 2019 Jul 8. PMID 31286262
- [Background] Ciocca L, Meneghello R, Monaco C, Savio G, Scheda L, Gatto MR, Baldissara P. In vitro assessment of the accuracy of digital impressions prepared using a single system for full-arch restorations on implants. Int J Comput Assist Radiol Surg. 2018 Jul;13(7):1097-1108. doi: 10.1007/s11548-018-1719-5. Epub 2018 Mar 2. PMID 29500759
- [Background] Chen Y, Zhai Z, Li H, Yamada S, Matsuoka T, Ono S, Nakano T. Influence of Liquid on the Tooth Surface on the Accuracy of Intraoral Scanners: An In Vitro Study. J Prosthodont. 2022 Jan;31(1):59-64. doi: 10.1111/jopr.13358. Epub 2021 May 29. PMID 33829613
- [Background] Carneiro Pereira AL, Medeiros VR, Campos MFTP, de Medeiros AKB, Yilmaz B, Carreiro ADFP. Conventional and digital impressions for complete-arch implant-supported fixed prostheses: time, implant quantity effect and patient satisfaction. J Adv Prosthodont. 2022 Aug;14(4):212-222. doi: 10.4047/jap.2022.14.4.212. Epub 2022 Aug 29. PMID 36105876
- [Background] Carbajal Mejia JB, Wakabayashi K, Nakamura T, Yatani H. Influence of abutment tooth geometry on the accuracy of conventional and digital methods of obtaining dental impressions. J Prosthet Dent. 2017 Sep;118(3):392-399. doi: 10.1016/j.prosdent.2016.10.021. Epub 2017 Feb 17. PMID 28222873
- [Background] Canullo L, Colombo M, Menini M, Sorge P, Pesce P. Trueness of Intraoral Scanners Considering Operator Experience and Three Different Implant Scenarios: A Preliminary Report. Int J Prosthodont. 2021 March/April;34(2):250-253. doi: 10.11607/ijp.6224. Epub 2020 Jun 26. PMID 32589002
- [Background] Arcuri L, Lio F, Campana V, Mazzetti V, Federici FR, Nardi A, Galli M. Influence of Implant Scanbody Wear on the Accuracy of Digital Impression for Complete-Arch: A Randomized In Vitro Trial. Materials (Basel). 2022 Jan 25;15(3):927. doi: 10.3390/ma15030927. PMID 35160873

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT05985226/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT05985226/ICF_001.pdf